CLINICAL TRIAL: NCT01554956
Title: A Historically Controlled Phase II/III Study to Evaluate Efficacy and Safety of Kedrion Human Plasminogen Eye Drop Preparation in Patients Diagnosed With Ligneous Conjunctivitis
Brief Title: Efficacy/Safety of Human Plasminogen Eye Drop in Ligneous Conjunctivitis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB046
Record Dates: First submitted 2011-12-20; First posted 2012-03-15 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-06

CONDITIONS: Ligneous Conjunctivitis
Keywords: Plasminogen Deficiency; Ligneous Conjunctivitis; Plasminogen; Ligneous Conjunctivitis in Plasminogen Deficient Patients
MeSH Terms: conditions — Plasminogen Deficiency, Type I; Congenital Plasminogen Deficiency | interventions — Plasminogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human Plasminogen (Experimental): Human Plasminogen Eye Drop treatment
  Interventions: Biological: Human Plasminogen

INTERVENTIONS:
Biological: Human Plasminogen — Eye Drops

SUMMARY:
Kedrion Human Plasminogen, a sterile human plasma-derived plasminogen preparation for topical ocular use will be evaluated for the indication of treatment of ligneous conjunctivitis.

KB046 will be an open-label, historically controlled clinical trial. At least 10 subjects with ligneous conjunctivitis, for approximately 20 eyes, will be treated and assessed. All subjects will receive the investigational medicinal product (IMP) for 12 to 48 weeks, with a possibility for extended treatment (Continuation segment)

DETAILED DESCRIPTION:
Kedrion Human Plasminogen, a sterile human plasma-derived plasminogen preparation for topical ocular use will be evaluated for the indication of treatment of ligneous conjunctivitis.

KB046 will be an open-label, historically controlled clinical trial. At least 10 subjects with ligneous conjunctivitis, for approximately 20 eyes, will be treated and assessed. All subjects will receive the investigational medicinal product (IMP) for 12 to 48 weeks, with a possibility for extended treatment (Continuation segment).

The study will be divided into 3 segments: segments 1 and 2 for assessment of efficacy and safety and segment 3 (continuation segment) assessing long-term safety. For each enrolled patient, both eyes will be treated regardless of unilateral or bilateral involvement. Treatment of the unaffected eyes provided data for the safety assessment. To assess efficacy, comparisons will be made against individual patient historical data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be diagnosed with ligneous conjunctivitis associated with Type I plasminogen deficiency, confirmed by the central laboratory and documented at pre-enrollment screening. The concomitant presence of other ligneous pseudomembranes at different sites will not constitute an exclusion criterion.
* Subjects should have documented historical records of disease course available for a period of at least 6 months surrounding an episode of LC, even if asymptomatic in the past for a newly diagnosed subject , including but not limited to age of LC onset, diagnosis of Plasminogen 1 deficiency, history of pseudomembrane lesions, disease duration, past treatment for LC, response to treatment and/or surgery (including regression and recurrence), before study entrance. If more history than 6 months surrounding an LC episode is available it will be included.
* Subjects, or their legally authorized representative, in the case of study participants < 18 years of age, should have been informed of the nature of the study, agreed to its provision, signed and dated the informed consent approved by the investigational review board (IRB) or ethics committee (EC).
* Subjects available for the duration of the study will be included. The Investigator will make sure that there is no plan for the subject to leave the area of the study site before the end of the study period. If they come from another center, they must agree to be compliant with the protocol mandated study visits and return for follow-up.

Exclusion Criteria:

* Subjects presenting ligneous conjunctivitis not associated with Type 1 plasminogen deficiency.
* Subjects with no history of LC lesions for Group 2, for Group 1 the entry lesions could be the first and included as history.
* Subject presenting antibodies against plasminogen at screening.
* Subjects with any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives, or participation in this trial.
* Subjects unwilling to give written informed consent or assent to participation.
* Subjects who have participated in another clinical trial within 1 month before study initiation, i.e. they have received any test drug within 30 days prior the study.
* Females of childbearing potential who are either pregnant or not using an adequate method of birth control
* Females who are breastfeeding.
* Subjects being treated with FFP or Laboratory Grade Plasminogen will undergo a washout period of at least 15 days before being considered for this study. This information will be disseminated to subjects ahead of their Screening Visit and will only occur following signing of the Informed Consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2014-04-25 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana, United States
- Italy (2):
  - Meyer Children's Hospital, Florence
  - AOU Padova, Padua

REFERENCES:
- [Derived] Caputo R, Shapiro AD, Sartori MT, Leonardi A, Jeng BH, Nakar C, Di Pasquale I, Price FW Jr, Thukral N, Suffredini AL, Pino L, Crea R, Mathew P, Calcinai M. Treatment of Ligneous Conjunctivitis with Plasminogen Eyedrops. Ophthalmology. 2022 Aug;129(8):955-957. doi: 10.1016/j.ophtha.2022.03.019. Epub 2022 Mar 26. No abstract available. PMID 35346720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 subjects were screened (11 in Part 1 and 2 in Part 2) of which 12 subjects (24 eyes) were enrolled in the study (11 in Part 1 and 1 in Part 2) and 1 subject who failed screening in Part 2. All subjects enrolled in Part 1 of the study were symptomatic at screening, so all were included in Group 1.
  No subjects were included in Group 2.
Pre-assignment Details: The study was divided in Part 1 (Segment 1 and Segment 2) and Part 2 (Continuation Segment). The screening procedures were performed within a 30-day window prior to receiving the first study IMP administration. A second screening for additional two subjects was performed before entering in the Part 2 of the study.
Units Other Than Participants: eyes
Groups:
- Group 1A: Symptomatic subjects with ocular pseudomembranes in one or both eyes at screening who received the IMP for 4 weeks (Segment 1) and with eyes showing complete pseudomembranes regression (defined as >90%). They have continued to received IMP at a reduced dose for an additional 8 weeks (Segment 2).
- Group 1B: Symptomatic subjects with ocular pseudomembranes in one or both eyes at screening who received the IMP for 4 weeks (Segment 1) and with eyes showing partial (defined as between 20% and 90%) or no pseudomembranes regression (defined as <20%). They were to undergo surgery, within 2 weeks from the end of Segment 1, to remove the pseudomembranes. After surgery, subjects were to continue receiving IMP for an additional 8 weeks, at the decreasing frequency.
- Continuation Segment: One additional patient, who entered directly in the Part 2, without previously completing the first part of the study and subjects demonstrating complete treatment success (defined as regression of pseudomembranes in Segment 1 and no relapse of pseudomembranes through Segment 2) at the end of the Segment 2 were entered the Continuation Segment.
Period: Part 1 (Segment 1 and Segment 2)
Arm/Group | Group 1A | Group 1B | Continuation Segment
Started | 4; 8 eyes (4 Symptomatic eyes (safety & efficacy evaluation) + 4 non symptomatic eyes (safety evaluation only)) | 7; 14 eyes (11 Symptomatic eyes (safety & efficacy evaluation) +3 non symptomatic eyes (safety evaluation only)) | 0; 0 eyes
Completed | 4; 8 eyes (4 Symptomatic eyes (safety & efficacy evaluation) + 4 non symptomatic eyes (safety evaluation only)) | 6; 12 eyes (9 Symptomatic eyes (safety & efficacy evaluation) +3 non symptomatic eyes (safety evaluation only)) | 0; 0 eyes
Not Completed | 0; 0 eyes | 1; 2 eyes | 0; 0 eyes
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Part 2 (Continuation Segment)
Arm/Group | Group 1A | Group 1B | Continuation Segment
Started | 4; 8 eyes | 6; 12 eyes | 1; 2 eyes (The total number of subjects enrolled in the trial was 12. According to study design 11 subjects were enrolled in the study Part 1. One subject dropped out and a total of 10 subjects completed the Part 1. All these 10 subjects entered in the study Part 2 and one additional subject was enrolled directly in this segment. Therefore a total of 11 subjects have been treated in the study Part 2.)
Completed | 2; 4 eyes | 1; 2 eyes | 0; 0 eyes
Not Completed | 2; 4 eyes | 5; 10 eyes | 1; 2 eyes
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — SUBJECT WAS WITHDRAWN BY THE INVESTIGATOR AT THE SITE FOR NON-IMP RELATED REASON | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Continuation Segment: Subjects demonstrating complete treatment success (defined as regression of pseudomembranes in Segment 1 and no relapse of pseudomembranes through Segment 2) at the end of the Segment 2 were entered the Continuation Segment and one additional patient, who entered directly in the Part 2, without previously completing the first part of the study.
- Total: Total of all reporting groups
Arm/Group | Group 1A | Group 1B | Continuation Segment | Total
Number analyzed (Participants) | 4 | 7 | 1 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 1 | 10
  Between 18 and 65 years | 1 | 1 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 0 | 7
  Male | 1 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 7 | 1 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Success to Prevent Pseudomembranes Relapse
Description: The primary endpoint (prevention of pseudomembrane relapse) was presented descriptively based on the predefined success levels: complete success (defined as no relapse by the end of Segment 2), partial success(defined as relapse appearing 2 weeks or longer after the start of Segment 2, or if following the 3 rd cycle of Segment 2 for Group 1A no relapse occurred while maintaining the higher dose) or failure (defined as relapse within 2 weeks of the start of Segment 2 or if at repeat cycles of Segment 1 for Group 1A, the pseudomembranes did not regress after Segment 1). Ninety-five percent confidence intervals for the relapse rate (complete success, and complete plus partial success) were calculated on the assumption of a binomial distribution. The responses were tabulated for the mITT and Per Protocol populations.
Time Frame: The prevention of pseudomembranes relapse was assessed during Segment 2, after initial total regression at the end of Segment 1 (Group 1A) or after surgical excision (Group 1B) up to 21 weeks from the study start.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: number of eyes
Groups:
- Group 1A_mITT: Modified ITT (mITT) population consists of all eyes of subjects assigned to Groups 1A at the start of Study Segment 2, who received at least one dose of the study treatment, and underwent at least one efficacy assessment in Segment 2
- Group 1B_mITT: Modified ITT (mITT) population consists of all eyes of subjects assigned to Group 1B at the start of Study Segment 2, who received at least one dose of the study treatment, and underwent at least one efficacy assessment in Segment 2
- Group 1A_PP: Per Protocol population consists of all eyes of Group 1A subjects included in the mITT population, who have completed both Segment 1 and Segment 2 of the study and received at least 80% of the protocol required doses of the study treatment without any major protocol violations or exceptions that could impact the integrity of study data.
- Group 1B_PP: Per Protocol population consists all eyes of Group 1B subjects included in the mITT population, who have completed both Segment 1 and Segment 2 of the study and received at least 80% of the protocol required doses of the study treatment without any major protocol violations or exceptions that could impact the integrity of study data.
Arm/Group | Group 1A_mITT | Group 1B_mITT | Group 1A_PP | Group 1B_PP
Number analyzed (Participants) | 4 | 7 | 3 | 6
Number analyzed (number of eyes) | 4 | 11 | 3 | 9
percentage of eyes
  success | 75 [19.4 to 99.4] | 81.8 [48.2 to 97.7] | 100 [29.2 to 100] | 100 [66.4 to 100]
  partial success | 0 [0 to 60.2] | 18.2 [2.3 to 51.8] | 0 [0 to 70.8] | 0 [0 to 33.6]
  failure | 25 [0.6 to 80.6] | 0 [0 to 28.5] | 0 [0 to 70.8] | 0 [0 to 33.6]

2. Secondary Outcome: Percentage of Eyes With Regression in Surface Area of Existing Ligneous Pseudomembranes
Description: The secondary endpoint was presented descriptively based on the predefined success levels: complete success (defined as regression of PSAs >90%), partial success (defined as regression of PSAs between 20% and 90%) or failure (defined as regression of PSAs <20%). The responses were tabulated for the mITT and the Per Protocol populations.
Time Frame: Regression of pseudomembranes surface area (PSA) was assessed from baseline to the end of Segment 1, up to 5 weeks (one subject was assessed after 9 weeks due to the occurrence of a not related SAE - Varicella - between Visit 0 and Visit 1)
Population: The first Part of the Study was divided in two segments: Segment 1, where all patients received the same intervention and Segment 2 where, depending on the outcome of Segment 1, patients were assigned to Group 1A (in case of complete pseudomembranes regression) or Group 1B (in case of no or partial pseudomembranes regression), receiving different intervention.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: number of eyes
Groups:
- Group 1_ mITT: mITT Population consists of all eyes assigned to Groups 1A and 1B at the start of study segment 2, who received at least one dose of the study treatment, and had at least one efficacy assessment in Segment 2.
- Group 1_PP: Per Protocol population includes all eyes of patients included in the mITT population, who have completed both Segment 1 and Segment 2 of the study and received at least 80% of the protocol required doses of the study treatment without any major protocol violations or exceptions that could impact the integrity of study data.
Arm/Group | Group 1_ mITT | Group 1_PP
Number analyzed (Participants) | 11 | 9
Number analyzed (number of eyes) | 15 | 12
percentage of eyes
  complete success | 20 [4.3 to 48.1] | 25 [5.5 to 57.2]
  partial success | 46.7 [21.3 to 73.4] | 58.3 [27.7 to 84.8]
  failure | 33.3 [11.8 to 61.6] | 16.7 [2.1 to 48.4]

3. Other Pre Specified Outcome: Number of Subjects Who Experience Signs and Symptoms of Sensitization.
Description: The safety parameters were presented descriptively and tabulated for the Group 1A, Group 1B and Continuation Segment safety population.
Time Frame: Signs and symptoms of sensitization were evaluated during the Part 1 and Part 2 of the study up to 7 years
Measure: Number; unit: number of subjects
Groups:
- Group 1A_Safety Population: Safety population consists of all Group 1A enrolled subjects who received at least one dose of the study treatment
- Group 1B_Safety Population: Safety population consists of all Group 1B enrolled subjects who received at least one dose of the study treatment
- Part 2 Continuation Segment_Safety Population: Safety population includes all subjects who received at least one dose of the study drug in the continuation segment period.
Arm/Group | Group 1A_Safety Population | Group 1B_Safety Population | Part 2 Continuation Segment_Safety Population
Number analyzed (Participants) | 4 | 7 | 11
number of subjects
  Number of Subjects with Ocular Adverse Events | 1 | 4 | 8
  Conjunctivitis bacterial | 1 | 0 | 2
  Ectropion | 0 | 1 | 0
  Eye haemorrhage | 0 | 1 | 0
  Eye pain | 0 | 1 | 1
  Eyelid margin crusting | 0 | 1 | 0
  Lacrimation increased | 0 | 1 | 0
  Ocular hyperaemia | 0 | 1 | 3
  Ocular hypertension | 0 | 1 | 2
  Blepharitis | 0 | 0 | 1
  Cataract | 0 | 0 | 1
  Chalazion | 0 | 0 | 1
  Conjunctival disorder | 0 | 0 | 1
  Conjunctival oedema | 0 | 0 | 2
  Conjunctivitis | 0 | 0 | 4
  Eye discharge | 0 | 0 | 3
  Eye swelling | 0 | 0 | 2
  Pinguecula | 0 | 0 | 1

4. Other Pre Specified Outcome: Number of Subjects Who Experience Adverse Events.
Description: as for outcome 3
Time Frame: AEs were collected from the screening visit and throughout the study up to 7 years
Measure: Number; unit: number of subjects
Arm/Group | Group 1A_Safety Population | Group 1B_Safety Population | Part 2 Continuation Segment_Safety Population
Number analyzed (Participants) | 4 | 7 | 11
number of subjects
  Number of Subjects with Adverse Events | 4 | 7 | 10
  Number of Subjects with Causally-Related Adverse Events | 0 | 3 | 6
  Number of Subjects Prematurely Withdrawn due to Adverse Events | 0 | 0 | 3
  Number of Subjects with Serious Adverse Events | 2 | 3 | 0
  Number of Subjects with Causally-Related Serious Adverse Events | 0 | 0 | 2

5. Other Pre Specified Outcome: Number of Subjects Who Develop Antibodies Against Bovine Aprotinin.
Description: as for outcome 3
Time Frame: The antibody development was detected during Part 1 and Part 2 of the study up to 7 years
Population: All participants enrolled in the study underwent to immunogenicity assessment. Participans in Part 1 was 11: 4 from Group 1A and 7 from Group 1B. Participants analysed in Part 2 was 11: 4 from Part 1-Group 1A, 6 from Part 1-Group 1B and 1 new patient enrolled directly in Part 2.
Measure: Number; unit: number of subjects
Groups:
- Part 1 - Group 1A_Safety Population: Safety population consists of all Group 1A enrolled subjects who received at least one dose of the study treatment
- Part 1 - Group 1B_Safety Population: Safety population consists of all Group 1B enrolled subjects who received at least one dose of the study treatment
- Part 2 - Continuation Segment_Safety Population: Safety population includes all subjects who received at least one dose of the study drug in the continuation segment period.
Arm/Group | Part 1 - Group 1A_Safety Population | Part 1 - Group 1B_Safety Population | Part 2 - Continuation Segment_Safety Population
Number analyzed (Participants) | 4 | 7 | 11
number of subjects
  New antibody development | 0 | 3 | 3
  Antibody Increasing | 0 | 1 | 0
  Antibody Decreasing | 0 | 1 | 0
  Antibody no changes | 0 | 1 | 0

6. Other Pre Specified Outcome: Number of Subjects Who Develop Antibodies Against Human Plasminogen.
Description: as for outcome 3
Time Frame: The antibody development was detected during the Part 1 and Part 2 of the study, up to 7 years
Measure: Number; unit: number of subjects
Groups:
- Continuation Segment_Safety Population: Safety population includes all subjects who received at least one dose of the study drug in the continuation segment period.
Arm/Group | Group 1A_Safety Population | Group 1B_Safety Population | Continuation Segment_Safety Population
Number analyzed (Participants) | 4 | 7 | 11
number of subjects | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs were collected from the screening visit and throughout the study up to 7 years
Description: AEs were collected by spontaneous reporting by the patient, by review of the Subject Diaries, and, during the visits at site, by asking the patient non-leading questions about how they felt since their last study visit
Groups:
- Group 1A: Patients with eyes showing complete pseudomembranes regression (defined as >90%) who have received IMP at a dose of 2 drops/eye 6 times/day for 8 weeks.
- Group 1B: Patients with eyes showing partial (defined as between 20% and 90%) or no pseudomembranes regression (defined as <20%) were to undergo surgery, within 2 weeks from the end of Segment 1, to remove the pseudomembranes. After surgery, patients were to continue receiving IMP (2 drops/eye) for an additional 8 weeks, at the decreasing frequency.
- Continuation Segment: Subjects demonstrating complete treatment success (defined as regression of pseudomembranes in Segment 1 and no relapse of pseudomembranes through Segment 2) at the end of part 1 and one additional patient, who entered directly, without previously completing the first part of the study were to receive IMP at a dosage regimen of 2 drops/eye 4 to 6 times/day at Investigator's discretion.
Arm/Group | Group 1A | Group 1B | Continuation Segment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/7 | 3/11
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1A (N=4) | Group 1B (N=7) | Continuation Segment (N=11)
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Drug specific antibody present (Investigations) | 0 | 1 | 1 — Anti-plasminogen antibody
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1A (N=4) | Group 1B (N=7) | Continuation Segment (N=11)
Hypertension (Vascular disorders) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Multiple allergies (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 3 | 7
Axillary pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 1
Cervix disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Genital labial adhesions (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Liver palpable subcostal (Investigations) | 1 | 0 | 0
Antibody test positive (Investigations) | 0 | 4 | 4
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2
Chalazion (Eye disorders) | 0 | 0 | 1
Conjunctivitis bacterial (Eye disorders) | 1 | 0 | 2
Ectropion (Eye disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 1
Eye pain (Eye disorders) | 0 | 1 | 1
Eyelid margin crusting (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 3
Ocular hypertension (Eye disorders) | 0 | 1 | 2
Blepharitis (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Conjunctival disorder (Eye disorders) | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 4
Eye discharge (Eye disorders) | 0 | 0 | 3
Eye swelling (Eye disorders) | 0 | 0 | 2
Pinguecula (Eye disorders) | 0 | 0 | 1
Conductive deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 3
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 2
Gingival oedema (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Teething (Gastrointestinal disorders) | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Subcutaneous haematoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Excoriation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Candida nappy rash (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 5
Nasopharyngitis (Infections and infestations) | 0 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1
Herpangina (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 4
Skin papilloma (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any results communication will be examined by the PIs and Sponsor 60 days before the submission. Sponsor should receive one copy of each publication proposed. The comments of Sponsor should be issued not beyond 60 days. PI cannot publish data which are considered to be common to such a study without the consent of the other PIs and previous review of Sponsor. In case of disagreement between the PIs, the the senior author and the Sponsor will discuss to find a common position.

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT01554956/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT01554956/SAP_001.pdf